CLINICAL TRIAL: NCT05437211
Title: Ability of a Virtual-reality Based Solution Aiming to Reduce Patient Burden Related to Repetitive Intravenous Perfusions. A Proof-of-concept Study in Hemophilia Patients Receiving Prophylactic Factor VIII or Factor IX Infusions
Brief Title: A Proof-of-concept Study to Reduce Treatment Burden in Haemophilia Participants Receiving Factor VIII and Factor IX Infusions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: TAK-660-4013; MACS-2020-120101 (Other: Takeda)
Record Dates: First submitted 2022-06-24; First posted 2022-06-29 (Actual); Results first posted 2025-06-05 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-05

CONDITIONS: Hemophilia
Keywords: Drug Therapy
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- VR-based Experimental Group (Experimental): Participants will receive Factor VIII or Factor IX infusion using a VR-based solution. The VR-based solution will be provided in a medical device CE marked and specifically developed by Deepsen, a French company specializing in e-health solutions to reduce pain. It includes both a mobile phone application (for an explanation on infusions) and a 3D mask to be used during infusions.
  Interventions: Device: Virtual-reality (VR) Based Solution

INTERVENTIONS:
Device: Virtual-reality (VR) Based Solution — VR-based solution comprises a mobile phone application including explanation on the different steps to be followed to perform infusions in satisfactory conditions, notably as regards safety, as well as VAS for pain and anxiety to be completed at each Factor VIII or Factor IX infusion between inclusion and the Week 4 visit. It also comprises a 3D mask (to be used before or during infusions) including simulation of the infusions themselves (before infusion) and a relaxing and distracting content (during and after infusions).

SUMMARY:
The main aim is to describe how the treatment burden and challenges of participants, relatives, and doctors during regular Factor VIII and Factor IX infusions to treat hemophilia evolve using a virtual-reality (VR) based solution. The study also aims to find out how well the VR based solution is tolerated and how satisfied the participants, relatives, and doctors are with it.

The VR-based solution includes a mobile phone app and a 3D mask.

Participants will use the VR-based solution while receiving prophylactic Factor VIII and Factor IX infusions for 4 weeks at home. Participants will visit the clinic for the last infusion; at this time data will be collected from participants, relatives, and doctors

ELIGIBILITY:
Inclusion criteria:

1. Male participant over the age of 6 years, with diagnosed Congenital Hemophilia A or B, whatever the severity is
2. Participant under long-term prophylaxis with intravenous Factor VIII or Factor IX infusions
3. Participant (or the legal guardians if participant age <18 years) able and willing to give written informed consent and to comply with the requirements of the study protocol
4. Participant affiliated to the national social security or beneficiary to such insurance

Exclusion criteria:

1. Participant with known or suspected hypersensitivity to virtual-reality based tools
2. Participant with central venous line for the administration of Factor VIII or Factor IX
3. Participant (and the legal guardians if participant age <18 years) with history of unreliability or non-cooperation (including for completion of self-reported questionnaires)
4. Participant (and the legal guardians if participant age <18 years) with insufficient comprehension of French language
5. Participant taking part in another clinical trial
6. Participant deprived of his liberty by judicial or administrative order

NB: participants with haemophilia A having participated in the test phase of the study could be included in the clinical study itself after a period of 4 months minimum with no use of the virtual-reality based solution.

Min Age: 6 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 24 (Actual)
Dates: Start 2023-06-23 (Actual); Primary Completion 2024-02-21 (Actual); Study Completion 2024-02-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (6):
- France (6):
  - Centre de Reference Hemophilie Unite D'Hemostase Clinique, Bron, Auvergne-Rhône-Alpes
  - CHU Estaing, Clermont-Ferrand, Auvergne-Rhône-Alpes
  - Hôpital de Hautepierre - Pôle MIRMED, Strasbourg, Grand Est
  - CHU Purpan, Toulouse, Haute-Garonne
  - CHU Pellegrin, Bordeaux, Nouvelle-Aquitaine
  - Hôpital Hôtel-Dieu, Nantes, Pays de la Loire Region

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/ For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link. — https://clinicaltrials.takeda.com/study-detail/dad25f4820fb4885?idFilter=%5B%22TAK-660-4013%22%5D

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at the 6 centres in France from 23 June 2023 to 21 February 2024.
Pre-assignment Details: A total of 24 male participants with Congenital Haemophilia A or B were enrolled in this study.
Groups:
- Virtual Reality (VR)-Based Experimental Group: With Autonomy: Haemophilia participants with autonomy received Factor VIII or Factor IX infusion using a VR-based solution for 4 weeks. The VR-based solution was a medical device Conformité Européene (CE) marked and specifically developed by Deepsen, a French company specializing in e-health solutions to reduce pain. It included both a mobile phone application (for an explanation on infusions) and a 3D mask to be used during infusions.
- VR-based Experimental Group: Without Autonomy: Haemophilia participants without autonomy received Factor VIII or Factor IX infusion using a VR-based solution for 4 weeks. The VR-based solution was provided in a medical device CE marked and specifically developed by Deepsen, a French company specializing in e-health solutions to reduce pain. It included both a mobile phone application (for an explanation on infusions) and a 3D mask to be used during infusions.
Period: Overall Study
Arm/Group | Virtual Reality (VR)-Based Experimental Group: With Autonomy | VR-based Experimental Group: Without Autonomy
Started | 14 | 10
Included Set (IS) (The IS included all eligible participants with or without assessment at the end of the Week 4 visit.) | 14 | 10
Full Analysis Set (FAS) (The FAS included all the participants of the IS for whose at least one assessment at the Week 4 visit was available.) | 13 | 9
Completed | 13 | 9
Not Completed | 1 | 1
Not completed — Patient's decision | 1 | 1

BASELINE CHARACTERISTICS:
Population: The IS included all eligible participants with or without assessment at the end of the Week 4 visit.
Groups:
- VR-based Experimental Group: With Autonomy: Haemophilia participants with autonomy received Factor VIII or Factor IX infusion using a VR-based solution for 4 weeks. The VR-based solution was a medical device CE marked and specifically developed by Deepsen, a French company specializing in e-health solutions to reduce pain. It included both a mobile phone application (for an explanation on infusions) and a 3D mask to be used during infusions.
- Total: Total of all reporting groups
Arm/Group | VR-based Experimental Group: With Autonomy | VR-based Experimental Group: Without Autonomy | Total
Number analyzed (Participants) | 14 | 10 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.3 (20.6) | 13.9 (10.6) | 28.7 (21.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 14 | 10 | 24
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Mean Absolute Values of Anxiety Measured by an Anxiety Visual Analogue Scale (A-VAS) Before Each Factor VIII or Factor IX Infusion in Participants and Caregivers
Description: The anxiety of participants and caregivers before each Factor VIII or Factor IX infusion was measured with a 10-points VAS. The A-VAS is a 10-centimeter (cm) line with anchor statements on the left (0:no anxiety) and on the right (10: extreme anxiety). An increase in score from 0 to 10 indicated a worsening of anxiety.
Time Frame: At Week 4
Population: The FAS included all the participants of the IS for whose at least one assessment at the Week 4 visit was available. Here, "number analyzed" signifies participants who were evaluable at specified timepoints for the categories.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | VR-based Experimental Group: With Autonomy | VR-based Experimental Group: Without Autonomy
Number analyzed (Participants) | 13 | 9
score on a scale
  A-VAS before infusion For Participants: number analyzed (Participants) | 4 | 0
  A-VAS before infusion For Participants | 0.2 (0.4) |
  A-VAS before infusion For Caregivers: number analyzed (Participants) | 9 | 9
  A-VAS before infusion For Caregivers | 1.5 (2.0) | 0.0 (0.0)

2. Primary Outcome: Number of Participants With Relative Variation in Anxiety Measured by an Anxiety Visual Analogue Scale (A-VAS) Before and After Each Factor VIII or Factor IX Infusion
Description: The anxiety of participants and caregivers before each Factor VIII or Factor IX infusion was measured with a 10-points VAS. The A-VAS is a 10 cm line with anchor statements on the left (0:no anxiety) and on the right (10: extreme anxiety). An increase in score from 0 to 10 indicated a worsening of anxiety. Participants are categorized based on their A-VAS score values at both Baseline (-5, -3, 0, and 9.1) and Week 4 (-5, -2.3, -1, 0 and 2). The A-VAS score reported within each category represent the mean difference between the score collected after and before infusion (after minus before). A negative value indicates an improvement in anxiety compared to the baseline score, while a positive value indicates a worsening of anxiety compared to the baseline score.
Time Frame: Baseline up to Week 4
Population: The FAS included all the participants of the IS for whose at least one assessment at the Week 4 visit was available. As per SAP, the data for this outcome measure were planned to be analyzed for pooled treatment groups (With Autonomy and Without Autonomy). Here, "number analyzed" signifies participants who were evaluable at specified timepoints for the categories.
Measure: Count of Participants; unit: Participants
Groups:
- Pooled Arm: VR-based Experimental Group: Participants received Factor VIII or Factor IX infusion using a VR-based solution. The VR-based solution was provided in a medical device CE marked and specifically developed by Deepsen, a French company specializing in e-health solutions to reduce pain. It included both a mobile phone application (for an explanation on infusions) and a 3D mask to be used during infusions.
Arm/Group | Pooled Arm: VR-based Experimental Group
Number analyzed (Participants) | 22
Participants
  Participants with variation of the anxiety VAS values between Baseline (-5) and Week 4 (-5): number analyzed (Participants) | 4
  Participants with variation of the anxiety VAS values between Baseline (-5) and Week 4 (-5) | 0
  Participants with variation of the anxiety VAS values between Baseline (-5) and Week 4 (-2.3): number analyzed (Participants) | 4
  Participants with variation of the anxiety VAS values between Baseline (-5) and Week 4 (-2.3) | 1
  Participants with variation of the anxiety VAS values between Baseline (-5) and Week 4 (-1): number analyzed (Participants) | 4
  Participants with variation of the anxiety VAS values between Baseline (-5) and Week 4 (-1) | 1
  Participants with variation of the anxiety VAS values between Baseline (-5) and Week 4 (0): number analyzed (Participants) | 4
  Participants with variation of the anxiety VAS values between Baseline (-5) and Week 4 (0) | 2
  Participants with variation of the anxiety VAS values between Baseline (-5) and Week 4 (2): number analyzed (Participants) | 4
  Participants with variation of the anxiety VAS values between Baseline (-5) and Week 4 (2) | 0
  Participants with variation of the anxiety VAS values between Baseline (-3) and Week 4 (-5): number analyzed (Participants) | 2
  Participants with variation of the anxiety VAS values between Baseline (-3) and Week 4 (-5) | 0
  Participants with variation of the anxiety VAS values between Baseline (-3) and Week 4 (-2.3): number analyzed (Participants) | 2
  Participants with variation of the anxiety VAS values between Baseline (-3) and Week 4 (-2.3) | 0
  Participants with variation of the anxiety VAS values between Baseline (-3) and Week 4 (-1): number analyzed (Participants) | 2
  Participants with variation of the anxiety VAS values between Baseline (-3) and Week 4 (-1) | 0
  Participants with variation of the anxiety VAS values between Baseline (-3) and Week 4 (0): number analyzed (Participants) | 2
  Participants with variation of the anxiety VAS values between Baseline (-3) and Week 4 (0) | 1
  Participants with variation of the anxiety VAS values between Baseline (-3) and Week 4 (2): number analyzed (Participants) | 2
  Participants with variation of the anxiety VAS values between Baseline (-3) and Week 4 (2) | 1
  Participants with variation of the anxiety VAS values between Baseline (0) and Week 4 (-5): number analyzed (Participants) | 15
  Participants with variation of the anxiety VAS values between Baseline (0) and Week 4 (-5) | 1
  Participants with variation of the anxiety VAS values between Baseline (0) and Week 4 (-2.3): number analyzed (Participants) | 15
  Participants with variation of the anxiety VAS values between Baseline (0) and Week 4 (-2.3) | 0
  Participants with variation of the anxiety VAS values between Baseline (0) and Week 4 (-1): number analyzed (Participants) | 15
  Participants with variation of the anxiety VAS values between Baseline (0) and Week 4 (-1) | 0
  Participants with variation of the anxiety VAS values between Baseline (0) and Week 4 (0): number analyzed (Participants) | 15
  Participants with variation of the anxiety VAS values between Baseline (0) and Week 4 (0) | 14
  Participants with variation of the anxiety VAS values between Baseline (0) and Week 4 (2): number analyzed (Participants) | 15
  Participants with variation of the anxiety VAS values between Baseline (0) and Week 4 (2) | 0
  Participants with variation of the anxiety VAS values between Baseline (9.1) and Week 4 (-5): number analyzed (Participants) | 1
  Participants with variation of the anxiety VAS values between Baseline (9.1) and Week 4 (-5) | 0
  Participants with variation of the anxiety VAS values between Baseline (9.1) and Week 4 (-2.3): number analyzed (Participants) | 1
  Participants with variation of the anxiety VAS values between Baseline (9.1) and Week 4 (-2.3) | 0
  Participants with variation of the anxiety VAS values between Baseline (9.1) and Week 4 (-1): number analyzed (Participants) | 1
  Participants with variation of the anxiety VAS values between Baseline (9.1) and Week 4 (-1) | 0
  Participants with variation of the anxiety VAS values between Baseline (9.1) and Week 4 (0): number analyzed (Participants) | 1
  Participants with variation of the anxiety VAS values between Baseline (9.1) and Week 4 (0) | 1
  Participants with variation of the anxiety VAS values between Baseline (9.1) and Week 4 (2): number analyzed (Participants) | 1
  Participants with variation of the anxiety VAS values between Baseline (9.1) and Week 4 (2) | 0

3. Primary Outcome: Number of Participants With Decrease of 2 Points Out of 10 Points in the A-VAS Scale Before Each Factor VIII or Factor IX Infusion
Description: The anxiety of participants and caregivers before each Factor VIII or Factor IX infusion was measured with a 10-points VAS. The A-VAS is a 10 cm line with anchor statements on the left (0:no anxiety) and on the right (10: extreme anxiety). An increase in score from 0 to 10 indicated a worsening of anxiety.
Time Frame: At Week 4
Population: The FAS included all the participants of the IS for whose at least one assessment at the Week 4 visit was available. As per SAP, the data for this outcome measure was planned to be analyzed for pooled treatment groups (With Autonomy and Without Autonomy).
Measure: Count of Participants; unit: Participants
Groups:
- Pooled Arm: VR-based Experimental Group: Haemophilia participants with autonomy or without autonomy received Factor VIII or Factor IX infusion using a VR-based solution for 4 weeks. The VR-based solution was a medical device CE marked and specifically developed by Deepsen, a French company specializing in e-health solutions to reduce pain. It included both a mobile phone application (for an explanation on infusions) and a 3D mask to be used during infusions.
Arm/Group | Pooled Arm: VR-based Experimental Group
Number analyzed (Participants) | 22
Participants | 5

4. Primary Outcome: Mean Absolute Values of the Pain Measured by a Pain Visual Analogue Scale (P-VAS) After Each Factor VIII or Factor IX Infusion in Participants
Description: The pain of participants after each Factor VIII or Factor IX infusion was measured with a 10-points VAS. The P-VAS is a 10 cm line with anchor statements on the left (0: no pain) and on the right (10: extreme pain). An increase in score from 0 to 10 indicated a worsening of pain.
Time Frame: At Week 4
Population: The FAS included all the participants of the IS for whose at least one assessment at the Week 4 visit was available.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | VR-based Experimental Group: With Autonomy | VR-based Experimental Group: Without Autonomy
Number analyzed (Participants) | 13 | 9
score on a scale | 1.4 (2.7) | 0.6 (1.7)

5. Primary Outcome: Number of Participants With Absolute Variation of the Pain Measured by a P-VAS Scale After Each Factor VIII or Factor IX Infusion
Description: The pain of participants after each Factor VIII or Factor IX infusion was measured with a 10-points VAS. The P-VAS is a 10 cm line with anchor statements on the left (0: no pain) and on the right (10: extreme pain). An increase in score from 0 to 10 indicated a worsening of pain. Participants are categorized based on P-VAS score values at both Baseline (0, 1.3, 2, 4 and 5) and Week 4 (0, 0.2, 0.4, 5 and 8). A positive value indicates worsening in pain compared to the baseline score.
Time Frame: Baseline up to Week 4
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Pooled Arm: VR-based Experimental Group
Number analyzed (Participants) | 22
Participants
  Participants with absolute variation of the P-VAS values between Baseline (0) and Week 4 (0): number analyzed (Participants) | 15
  Participants with absolute variation of the P-VAS values between Baseline (0) and Week 4 (0) | 13
  Participants with absolute variation of the P-VAS values between Baseline (0) and Week 4 (0.2): number analyzed (Participants) | 15
  Participants with absolute variation of the P-VAS values between Baseline (0) and Week 4 (0.2) | 0
  Participants with absolute variation of the P-VAS values between Baseline (0) and Week 4 (0.4): number analyzed (Participants) | 15
  Participants with absolute variation of the P-VAS values between Baseline (0) and Week 4 (0.4) | 0
  Participants with absolute variation of the P-VAS values between Baseline (0) and Week 4 (5): number analyzed (Participants) | 15
  Participants with absolute variation of the P-VAS values between Baseline (0) and Week 4 (5) | 1
  Participants with absolute variation of the P-VAS values Baseline (0) and Week 4 (8): number analyzed (Participants) | 15
  Participants with absolute variation of the P-VAS values Baseline (0) and Week 4 (8) | 1
  Participants with absolute variation of the P-VAS values between Baseline (1.3) and Week 4 (0): number analyzed (Participants) | 1
  Participants with absolute variation of the P-VAS values between Baseline (1.3) and Week 4 (0) | 1
  Participants with absolute variation of the P-VAS values between Baseline (1.3) and Week 4 (0.2): number analyzed (Participants) | 1
  Participants with absolute variation of the P-VAS values between Baseline (1.3) and Week 4 (0.2) | 0
  Participants with absolute variation of the P-VAS values between Baseline (1.3) and Week 4 (0.4): number analyzed (Participants) | 1
  Participants with absolute variation of the P-VAS values between Baseline (1.3) and Week 4 (0.4) | 0
  Participants with absolute variation of the P-VAS values between Baseline (1.3) and Week 4 (5): number analyzed (Participants) | 1
  Participants with absolute variation of the P-VAS values between Baseline (1.3) and Week 4 (5) | 0
  Participants with absolute variation of the P-VAS values between Baseline (1.3) and Week 4 (8): number analyzed (Participants) | 1
  Participants with absolute variation of the P-VAS values between Baseline (1.3) and Week 4 (8) | 0
  Participants with absolute variation of the P-VAS values between Baseline (2) and Week 4 (0): number analyzed (Participants) | 1
  Participants with absolute variation of the P-VAS values between Baseline (2) and Week 4 (0) | 0
  Participants with absolute variation of the P-VAS values between Baseline (2) and Week 4 (0.2): number analyzed (Participants) | 1
  Participants with absolute variation of the P-VAS values between Baseline (2) and Week 4 (0.2) | 0
  Participants with absolute variation of the P-VAS values between Baseline (2) and Week 4 (0.4): number analyzed (Participants) | 1
  Participants with absolute variation of the P-VAS values between Baseline (2) and Week 4 (0.4) | 0
  Participants with absolute variation of the P-VAS values between Baseline (2) and Week 4 (5): number analyzed (Participants) | 1
  Participants with absolute variation of the P-VAS values between Baseline (2) and Week 4 (5) | 1
  Participants with absolute variation of the P-VAS values between Baseline (2) and Week 4 (8): number analyzed (Participants) | 1
  Participants with absolute variation of the P-VAS values between Baseline (2) and Week 4 (8) | 0
  Participants with absolute variation of the P-VAS values between Baseline (4) and Week 4 (0): number analyzed (Participants) | 2
  Participants with absolute variation of the P-VAS values between Baseline (4) and Week 4 (0) | 2
  Participants with absolute variation of the P-VAS values between Baseline (4) and Week 4 (0.2): number analyzed (Participants) | 2
  Participants with absolute variation of the P-VAS values between Baseline (4) and Week 4 (0.2) | 0
  Participants with absolute variation of the P-VAS values between Baseline (4) and Week 4 (0.4): number analyzed (Participants) | 2
  Participants with absolute variation of the P-VAS values between Baseline (4) and Week 4 (0.4) | 0
  Participants with absolute variation of the P-VAS values between Baseline (4) and Week 4 (5): number analyzed (Participants) | 2
  Participants with absolute variation of the P-VAS values between Baseline (4) and Week 4 (5) | 0
  Participants with absolute variation of the P-VAS values between Baseline (4) and Week 4 (8): number analyzed (Participants) | 2
  Participants with absolute variation of the P-VAS values between Baseline (4) and Week 4 (8) | 0
  Participants with absolute variation of the P-VAS values between Baseline (5) and Week 4 (0): number analyzed (Participants) | 3
  Participants with absolute variation of the P-VAS values between Baseline (5) and Week 4 (0) | 0
  Participants with absolute variation of the P-VAS values between Baseline (5) and Week 4 (0.2): number analyzed (Participants) | 3
  Participants with absolute variation of the P-VAS values between Baseline (5) and Week 4 (0.2) | 1
  Participants with absolute variation of the P-VAS values between Baseline (5) and Week 4 (0.4): number analyzed (Participants) | 3
  Participants with absolute variation of the P-VAS values between Baseline (5) and Week 4 (0.4) | 1
  Participants with absolute variation of the P-VAS values between Baseline (5) and Week 4 (5): number analyzed (Participants) | 3
  Participants with absolute variation of the P-VAS values between Baseline (5) and Week 4 (5) | 1
  Participants with absolute variation of the P-VAS values between Baseline (5) and Week 4 (8): number analyzed (Participants) | 3
  Participants with absolute variation of the P-VAS values between Baseline (5) and Week 4 (8) | 0

6. Primary Outcome: Number of Participants With a Decrease of 2 Points Out of 10 Points in the P-VAS Scale After Each Factor VIII or Factor IX Infusion
Description: as for outcome 4
Time Frame: Baseline up to Week 4
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Pooled Arm: VR-based Experimental Group
Number analyzed (Participants) | 22
Participants | 4

7. Primary Outcome: Mean Absolute Values of Anxiety Measured by an A-VAS Scale After Each Factor VIII or Factor IX Infusion in Participants and Caregivers
Description: as for outcome 3
Time Frame: At Week 4
Population: The FAS included all the participants of the IS for whose at least one assessment at the Week 4 visit was available. Here, "overall number of participants analyzed" signifies participants who were evaluable for this outcome measure and "number analyzed" signifies participants who were evaluable at specified timepoints.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | VR-based Experimental Group: With Autonomy | VR-based Experimental Group: Without Autonomy
Number analyzed (Participants) | 9 | 9
score on a scale
  A-VAS after infusion for participants: number analyzed (Participants) | 4 | 0
  A-VAS after infusion for participants | 0.2 (0.4) |
  A-VAS after infusion for caregivers | 0.8 (2.0) | 0.0 (0.0)

8. Primary Outcome: Number of Participants With a Decrease of 2 Points Out of 10 Points in the A-VAS Scale After Each Factor VIII or Factor IX Infusion
Description: The anxiety of participants and caregivers before each Factor VIII or Factor IX infusion was measured with a 10-points VAS. The A-VAS is a 10 cm line with anchor statements on the left (0:no anxiety) and on the right (10: extreme anxiety). An increase in score from 0 to 10 indicated a worsening of anxiety and negative value indicated worst health.
Time Frame: Baseline up to Week 4
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Pooled Arm: VR-based Experimental Group
Number analyzed (Participants) | 22
Participants | 2

9. Primary Outcome: Absolute Variation of Caregivers and Adult Participants Quality of Life Measured With the European Quality of Life 5 Dimensions 3-Levels (EQ-5D-3L) Health State Index Score
Description: The EQ-5D-3L is a standardized instrument for use as a measure of health outcome and was administered to adult participants to assess the effect of the treatment on the participants' quality of life. Adult participants selected answer for each of the following 3-level dimensions: 1) mobility; 2) self-care; 3) usual activities; 4) pain/discomfort; 5) anxiety/depression used to compute an index score ranging from 0 (worst imaginable health state) to 1 (best imaginable health state). An increase in the EQ-5D-3L index score indicated improvement and negative value indicated worst health.
Time Frame: At Week 4
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | VR-based Experimental Group: With Autonomy | VR-based Experimental Group: Without Autonomy
Number analyzed (Participants) | 9 | 5
score on a scale
  Absolute Variation for adult participants: number analyzed (Participants) | 9 | 2
  Absolute Variation for adult participants | 0.0 (0.2) | -0.0 (0.1)
  Absolute Variation for caregivers: number analyzed (Participants) | 2 | 5
  Absolute Variation for caregivers | 0.3 (0.1) | -0.0 (0.1)

10. Primary Outcome: Relative Variation of Caregivers and Adult Participants Quality of Life Measured With the European Quality of Life 5 Dimensions 3-Levels (EQ-5D-3L) Health State Index Score
Description: The EQ-5D-3L is a standardized instrument for use as a measure of health outcome and was administered to adult participants to assess the effect of the treatment on the participants' quality of life. Adult participants selected answer for each of the following 3-level dimensions: 1) mobility; 2) self-care; 3) usual activities; 4) pain/discomfort; 5) anxiety/depression used to compute an index score ranging from 0 (worst imaginable health state) to 1 (best imaginable health state). An increase in the EQ-5D-3L index score indicated improvement and negative value indicated worst health. Relative variation from baseline at visit (%) = 100 * Absolute change from baseline at visit (in units) / value at baseline (in units).
Time Frame: At Week 4
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | VR-based Experimental Group: With Autonomy | VR-based Experimental Group: Without Autonomy
Number analyzed (Participants) | 9 | 5
percentage
  Relative Variation for adult participants: number analyzed (Participants) | 9 | 2
  Relative Variation for adult participants | 7.1 (32.7) | -5.1 (7.2)
  Relative Variation for caregivers: number analyzed (Participants) | 2 | 5
  Relative Variation for caregivers | 61.0 (34.8) | -2.0 (11.8)

11. Primary Outcome: Absolute Variation of Youth Participants Quality of Life Measured With the European Quality of Life 5 Dimensions For Youth (EQ-5D-Y) Health State Index Score
Description: The EQ-5D-Y is a standardized instrument for use as a measure of health outcome and was administered to youth participants to assess the effect of the treatment on the participants' quality of life. Youth participants selected answer for each of the following 3-level dimensions: 1) mobility; 2) self-care; 3) usual activities; 4) pain/discomfort; 5) anxiety/depression used to compute an index score ranging from 0 (worst imaginable health state) to 1 (best imaginable health state). An increase in the EQ-5D-Y index score indicated improvement and negative value indicated worst health.
Time Frame: At Week 4
Population: The FAS included all the participants of the IS for whose at least one assessment at the Week 4 visit was available. Here" overall number of participants analyzed" signifies participants who were evaluable for this outcome measure and" number analyzed" signifies participants who were evaluable at specified timepoints.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | VR-based Experimental Group: With Autonomy | VR-based Experimental Group: Without Autonomy
Number analyzed (Participants) | 4 | 7
score on a scale | -0.1 (0.2) | -0.1 (0.3)

12. Primary Outcome: Relative Variation of Youth Participants Quality of Life Measured With the European Quality of Life 5 Dimensions For Youth (EQ-5D-Y) Health State Index Score
Description: The EQ-5D-Y is a standardized instrument for use as a measure of health outcome and was administered to youth participants to assess the effect of the treatment on the participants' quality of life. Youth participants selected answer for each of the following 3-level dimensions: 1) mobility; 2) self-care; 3) usual activities; 4) pain/discomfort; 5) anxiety/depression used to compute an index score ranging from 0 (worst imaginable health state) to 1 (best imaginable health state). An increase in the EQ-5D-Y index score indicated improvement and negative value indicated worst health. Relative variation from baseline at visit (%) = 100 * Absolute change from baseline at visit (in units) / value at baseline (in units).
Time Frame: At Week 4
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | VR-based Experimental Group: With Autonomy | VR-based Experimental Group: Without Autonomy
Number analyzed (Participants) | 4 | 7
percentage | -21.2 (35.3) | -12.8 (32.8)

13. Primary Outcome: Number of Participants and Caregivers With a Decrease of 2 Points in the EQ-5D-3L VAS and EQ-5D-Y Score
Description: EQ-5D-3L health questionnaire is adult participant and caregivers and EQ-5D-Y is a youth participant answered questionnaire scoring 5 dimensions - mobility, self-care, usual activities, pain/discomfort and anxiety/depression. The status of each dimension had 3 possible responses (1 =no problem, 2 =some problem 3 =extreme problems) in the relevant health dimension. Higher score indicated a worsening health condition.
Time Frame: At Week 4
Population: The FAS included all the participants of the IS for whose at least one assessment at the Week 4 visit was available. Here, "number analyzed" signifies participants who were evaluable at specified timepoints.
Measure: Count of Participants; unit: Participants
Arm/Group | Virtual Reality (VR)-Based Experimental Group: With Autonomy | VR-based Experimental Group: Without Autonomy
Number analyzed (Participants) | 13 | 9
Participants
  EQ-5D-3L Score for Participants | 0 | 0
  EQ-5D-3L Score for Caregivers | 0 | 0
  EQ-5D-Y Score for Youth Participants | 0 | 0

14. Primary Outcome: Absolute Variation of All Participants Anxiety Measured by State-Trait Anxiety Inventory (STAI-Y) Score
Description: The STAI is a psychological inventory consisting of 40 self-report items on a 4-point Likert scale. The STAI measures two types of anxiety - state anxiety (STAI-Y1) and trait anxiety (STAI-Y2). Higher scores were positively correlated with higher levels of anxiety. Each type of anxiety has its own scale of 20 different questions and were rated on a 4-point scale (e.g. from 'Almost Never to 'Almost Always'). Low scores indicated a mild form of anxiety, and high scores indicated a severe form of anxiety. STAI score ranged from 20 to 80 where higher scores indicated greater anxiety and negative value indicated worst anxiety.
Time Frame: At Week 4
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | VR-based Experimental Group: With Autonomy | VR-based Experimental Group: Without Autonomy
Number analyzed (Participants) | 13 | 9
Score on a scale
  Absolute variation of the STAI-Y1 | -2.4 (7.2) | -1.5 (3.9)
  Absolute variation of the STAI-Y2: number analyzed (Participants) | 12 | 9
  Absolute variation of the STAI-Y2 | -2.9 (3.1) | -0.5 (3.0)

15. Primary Outcome: Relative Variation of All Participants Anxiety Measured by State-Trait Anxiety Inventory (STAI-Y) Score
Description: The STAI is a psychological inventory consisting of 40 self-report items on a 4-point Likert scale. The STAI measures two types of anxiety - state anxiety (STAI-Y1) and trait anxiety (STAI-Y2). Higher scores were positively correlated with higher levels of anxiety. Each type of anxiety has its own scale of 20 different questions and were rated on a 4-point scale (e.g. from 'Almost Never to 'Almost Always'). Low scores indicated a mild form of anxiety, and high scores indicated a severe form of anxiety. STAI score ranged from 20 to 80 where higher scores indicated greater anxiety and negative value indicated worst anxiety. Relative variation from baseline at visit (%) = 100 * Absolute change from baseline at visit (in units) / value at baseline (in units).
Time Frame: At Week 4
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | VR-based Experimental Group: With Autonomy | VR-based Experimental Group: Without Autonomy
Number analyzed (Participants) | 13 | 9
percentage
  Relative variation of the STAI-Y1 | -6.6 (21.0) | -3.7 (12.7)
  Relative variation of the STAI-Y2: number analyzed (Participants) | 12 | 9
  Relative variation of the STAI-Y2 | -8.1 (8.1) | -1.5 (10.2)

16. Primary Outcome: Number of All Participants With Decrease of at Least One Level of State-Trait Anxiety Inventory Severity (STAI-S)
Description: The STAI-S is a psychological assessment tool used to measure the level of anxiety a person is experiencing at a particular moment in time that assesses both State anxiety (STAI-Y1) and Trait anxiety (STAI-Y2). Each type of anxiety has its own scale of 20 different questions each that are scored on a 4-point scale evaluating how respondents feel "right now, at this moment" (e.g. from 'Almost Never to 'Almost Always'). Total scores for each (Y1 and Y2) range from 20 to 80, with higher scores correlating with greater anxiety. Severity for each STAI-Y1 and STAI-Y2 is defined by the scores on STAI-S: 20-35 (very low) 36-45 (low) 46-55 (moderate) 56-65 (high) 66-80 (very high). Number of participants with decrease of at least one level of State-Trait Anxiety Inventory- Severity (STAI-S) are reported.
Time Frame: At Week 4
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | VR-based Experimental Group: With Autonomy | VR-based Experimental Group: Without Autonomy
Number analyzed (Participants) | 13 | 9
Participants
  Decrease from baseline of at least one level of anxiety state of STAI-Y1 | 3 | 2
  Decrease from baseline of at least one level of anxiety state of STAI-Y2: number analyzed (Participants) | 12 | 9
  Decrease from baseline of at least one level of anxiety state of STAI-Y2 | 4 | 1

17. Primary Outcome: Absolute Variation of Participants Depression Measured by Patient Health Questionnaire (Module 9) (PHQ-9) Depression Severity
Description: The PHQ-9 measures self-reports of depressive symptoms within the prior 2 weeks and has been well-validated, shown high test-retest reliability, shown high internal consistency, and shown to be responsive to changes in treatment. Response options were on a 4-point scale (0 = not at all, 3 = nearly every day). The overall PHQ-9 score ranged from 0 to 27 where 0-5 (none) 5-10 (mild) 10-15 (moderate) 15-20 (moderately severe) 20-27 (severe). Higher values represented more severe depression status.
Time Frame: At Week 4
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | VR-based Experimental Group: With Autonomy | VR-based Experimental Group: Without Autonomy
Number analyzed (Participants) | 13 | 8
score on a scale | -1.3 (3.2) | -1.4 (4.9)

18. Primary Outcome: Relative Variation of Participants Depression Measured by Patient Health Questionnaire (Module 9) (PHQ-9) Depression Severity
Description: The PHQ-9 measures self-reports of depressive symptoms within the prior 2 weeks and has been well-validated, shown high test-retest reliability, shown high internal consistency, and shown to be responsive to changes in treatment. Response options were on a 4-point scale (0 = not at all, 3 = nearly every day). The overall PHQ-9 score ranged from 0 to 27 where 0-5 (none) 5-10 (mild) 10-15 (moderate) 15-20 (moderately severe) 20-27 (severe). Higher values represented more severe depression status. Relative variation from baseline at visit (%) = 100 * Absolute change from baseline at visit (in units) / value at baseline (in units).
Time Frame: At Week 4
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | VR-based Experimental Group: With Autonomy | VR-based Experimental Group: Without Autonomy
Number analyzed (Participants) | 12 | 7
percentage | -13.7 (28.2) | 51.9 (161.2)

19. Primary Outcome: Number of Participants With Decrease of at Least One Level of Depression Severity Measured by PHQ-9 Scale
Description: as for outcome 17
Time Frame: Baseline up to Week 4
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | VR-based Experimental Group: With Autonomy | VR-based Experimental Group: Without Autonomy
Number analyzed (Participants) | 13 | 8
Participants | 2 | 3

20. Primary Outcome: Number of Participants With Absolute Adherence to Infusions Measured by 4-Item Morisky Medication Adherence Scale (MMAS-4) Scores
Description: The Morisky Medication Adherence Scale in the original version (MMAS-4) is a structured self-report measure of medication-taking behaviour. It consisted of 4 items, with binary scoring (yes/no). Participants scored one point for every 'Yes' answer. A score of 0 to 1 indicated low adherence; a score of 2 to 3 indicated medium adherence, and a score of 4 indicated high adherence.
Time Frame: Baseline up to Week 4
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | VR-based Experimental Group: With Autonomy | VR-based Experimental Group: Without Autonomy
Number analyzed (Participants) | 13 | 9
Participants | 7 | 6

21. Primary Outcome: Number of Participants With Changes in Adherence to Infusions Measured by MMAS-4 by Classes
Description: as for outcome 20
Time Frame: Baseline up to Week 4
Population: The FAS included all the participants of the IS for whose at least one assessment at the Week 4 visit was available.
Measure: Count of Participants; unit: Participants
Arm/Group | VR-based Experimental Group: With Autonomy | VR-based Experimental Group: Without Autonomy
Number analyzed (Participants) | 13 | 9
Participants
  Participants with changes in Low adherence (0-1) | 0 | 0
  Participants with changes in Medium adherence (2-3) | 6 | 3
  Participants with changes in High adherence (4) | 7 | 6

22. Primary Outcome: Number of Participants Who Scored 4 (High Adherence) Using MMAS-4 Scale at Week 4
Description: The Morisky Medication Adherence Scale in the original version (MMAS-4) is a structured self-report measure of medication-taking behavior. It consisted of 4 items, with binary scoring (yes/no). Participants scored one point for every 'Yes' answer. A score of 0 to 1 indicated low adherence; a score of 2 to 3 indicated medium adherence, and a score of 4 indicated high adherence.
Time Frame: At Week 4
Population: The FAS included all the participants of the IS for whose at least one assessment at the Week 4 visit was available.
Measure: Count of Participants; unit: Participants
Arm/Group | VR-based Experimental Group: With Autonomy | VR-based Experimental Group: Without Autonomy
Number analyzed (Participants) | 13 | 9
Participants | 7 | 6

23. Primary Outcome: Number of Participants and Caregivers With Adherence to VR-Based Solutions at Week 4
Description: Adherence to the VR-based solution was assessed at Week 4 using the MMAS. The Morisky Medication Adherence Scale in the original version (MMAS-4) is a structured self-report measure of medication-taking behaviour. It consisted of 4 items, with binary scoring (yes/no). Participants scored one point for every 'Yes' answer. A score of 0 to 1 indicated low adherence; a score of 2 to 3 indicated medium adherence, and a score of 4 indicated high adherence.
Time Frame: At Week 4
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | VR-based Experimental Group: With Autonomy | VR-based Experimental Group: Without Autonomy
Number analyzed (Participants) | 13 | 9
Participants
  Participants with Low adherence (0-1) | 1 | 0
  Participants with Medium adherence (2-3) | 6 | 5
  Participants with High adherence (4) | 6 | 4
  Caregivers with Low adherence (0-1): number analyzed (Participants) | 3 | 5
  Caregivers with Low adherence (0-1) | 0 | 0
  Caregivers with Medium adherence (2-3): number analyzed (Participants) | 3 | 5
  Caregivers with Medium adherence (2-3) | 2 | 0
  Caregivers with High adherence (4): number analyzed (Participants) | 3 | 5
  Caregivers with High adherence (4) | 1 | 5

24. Primary Outcome: Number of Participants With a Patients' Global Impression of Change (PGIC) Score Greater Than (>) 3 Among Participants and Caregivers
Description: The PGIC is a 7-point Likert scale, a verbal rating scale that asked the respondent to best describe change in symptoms compared to the beginning of study. Participants/caregivers selected from scale range of 1 (very much worsened) to 7 (very much improved). Higher score indicated improved outcome.
Time Frame: At Week 4
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | VR-based Experimental Group: With Autonomy | VR-based Experimental Group: Without Autonomy
Number analyzed (Participants) | 13 | 9
Participants
  PGIC: Patients (Score >3) | 7 | 4
  PGIC: Caregivers (Score >3): number analyzed (Participants) | 3 | 5
  PGIC: Caregivers (Score >3) | 2 | 2

25. Secondary Outcome: Number of Participants, With Satisfaction, Willingness to Continue the VR-Based Solution Measured by 4-point Likert Scale Score More Than and Equal to (>=3) Among Participants and Caregivers
Description: A 4-point Likert scale was used to assess the number of participants, caregivers, and investigators with a score of 3 or 4 (satisfied or very satisfied) with the use of the VR- based system. The Likert scale is composed from 1=never satisfied to 4=very satisfied.
Time Frame: At Week 4
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | VR-based Experimental Group: With Autonomy | VR-based Experimental Group: Without Autonomy
Number analyzed (Participants) | 13 | 9
Participants
  Satisfaction: Participants (Score >=3) | 10 | 9
  Satisfaction: Caregivers (Score >=3): number analyzed (Participants) | 3 | 5
  Satisfaction: Caregivers (Score >=3) | 2 | 4

26. Secondary Outcome: Number of Participants With Preference and No-preference for the VR-Based Solution Using a Binary Question Among Participants and Caregivers
Description: Preference for the VR-based solution in participants and caregivers was assessed using a binary question: Yes (Preference for the VR-based solution) and No (preference for VR-based solution) was assessed.
Time Frame: At Week 4
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | VR-based Experimental Group: With Autonomy | VR-based Experimental Group: Without Autonomy
Number analyzed (Participants) | 13 | 9
Participants
  Preference for the VR-based solution - Participants: Yes | 5 | 7
  Preference for the VR-based solution - Participants: No | 8 | 2
  Preference for the VR-based solution - Caregivers: number analyzed (Participants) | 3 | 5
  Preference for the VR-based solution - Caregivers: Yes | 2 | 4
  Preference for the VR-based solution - Caregivers: No | 1 | 1

27. Secondary Outcome: Number of Incidents With the VR-Based Solution
Description: An incident is a minor hardware and/or software event that prevents the correct use of the solution in its context. The incidents were mainly associated with misuse by the user of the solution or with a software and/or hardware failure.
Time Frame: Baseline up to Week 4
Population: The IS included all eligible participants with or without assessment at the end of the Week 4 visit.
Measure: Number; unit: number of incidents
Arm/Group | VR-based Experimental Group: With Autonomy | VR-based Experimental Group: Without Autonomy
Number analyzed (Participants) | 14 | 10
number of incidents | 3 | 1

28. Secondary Outcome: Number of Participants With Related Adverse Events (AEs) and Serious Adverse Events (SAEs) to the Infusions of Factor VIII or Factor IX or VR-Based Solution
Description: An AE is any untoward medical occurrence in a participant administered a medicinal product and which does not necessarily have to have a causal relationship with this treatment. AEs related to infusions of Factor VIII or Factor IX or use of VR-based solution was assessed. An SAE is any untoward medical occurrence that at any dose: results in death, is a life-threatening event, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, results in a congenital anomaly/birth defect or any other medically important event that, in the opinion of the healthcare provider, may jeopardize the participant or may require intervention to prevent one of the other outcomes listed in the definition above.
Time Frame: From start of study up to Week 4
Population: The IS included all eligible participants with or without assessment at the end of the Week 4 visit.
Measure: Count of Participants; unit: Participants
Arm/Group | VR-based Experimental Group: With Autonomy | VR-based Experimental Group: Without Autonomy
Number analyzed (Participants) | 14 | 10
Participants
  Participants with related AEs | 0 | 0
  Participants with SAEs | 0 | 0

ADVERSE EVENTS:
Time Frame: From start of study up to Week 4
Description: The IS included all eligible participants with or without assessment at the end of the Week 4 visit.
Arm/Group | VR-based Experimental Group: With Autonomy | VR-based Experimental Group: Without Autonomy
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/10
Other Adverse Events (participants affected / at risk) | 2/14 | 0/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | VR-based Experimental Group: With Autonomy (N=14) | VR-based Experimental Group: Without Autonomy (N=10)
Headache (Nervous system disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2023-02-28): https://cdn.clinicaltrials.gov/large-docs/11/NCT05437211/Prot_000.pdf
  • Statistical Analysis Plan (2024-05-14): https://cdn.clinicaltrials.gov/large-docs/11/NCT05437211/SAP_001.pdf